CLINICAL TRIAL: NCT01224379
Title: Clinical Trial of the Efficacy of Hybrid Systems(Topping Off)in Comparison to the Conventional Spondylodesis in Fusion-surgery in the Lumbal Spine: a Prospective, Randomised Study
Brief Title: Comparison of Standard Fusion With "Topping Off"-System in Lumbar Spine
Acronym: Topping-off
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Cologne (Other)
Responsible Party: University of Cologne, Medizinische Fakultät der Universität zu Köln
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Uni-Köln-1223; Uni-Köln-1223 (Other Grant/Funding Number: University of Cologne)
Record Dates: First submitted 2010-10-19; First posted 2010-10-20 (Estimated); Last update posted 2010-10-20 (Estimated); Status verified 2010-09

CONDITIONS: Spondylolisthesis; Erosive Osteochondrosis in L2-S1
Keywords: Lumbar spine; fusion; adjacent instability; topping-off.
MeSH Terms: conditions — Spondylolisthesis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm1: "topping off" system (Other): The intervention group will receive a "topping off" system (PLIF -posterior intervertebral fusion- connected with a flexible pedicle screw system above the fusion).
  Interventions: Device: Topping off system
- Arm 2: monosegmental PLIF (Other): The control group receives a monosegmental PLIF. This is the current standard therapy for many pathologies in the lumbar spine (e.g. Spondylolisthesis)
  Interventions: Device: monosegmental PLIF

INTERVENTIONS:
Device: Topping off system — The intervention group will receive a "topping off" system (PLIF -posterior intervertebral fusion- connected with a flexible pedicle screw system above the fusion).
  Other Names: Topping off
  Arms: Arm1: "topping off" system
Device: monosegmental PLIF — The control group receives a monosegmental PLIF. This is the current standard therapy for many pathologies in the lumbar spine (e.g. Spondylolisthesis)
  Arms: Arm 2: monosegmental PLIF

SUMMARY:
Does a new "topping-off" device lead to a better clinical outcome compared to standard fusion? Does this device prevent the development of adjacent instability? Does radiological adjacent instability correlate with clinical outcome?

DETAILED DESCRIPTION:
Primary efficacy endpoint:

The baseline and follow-up values after 6 weeks after the operation as well as 6 and 12 months after baseline of the SF-36 (Short-Form-36)-Measured Outcome regarding the Physical Component Summary (PCS).

Key secondary endpoint(s):

1. Mental Component Summary (MCS) and individual dimensions and subscales of the SF-36
2. Individual dimensions of the Oswestry Disability Index (ODI)
3. Time until radiological adjacent instability and comparison to the clinical outcome
4. Capacity of work at the time of surgery and after surgery, time until return to work

Assessment of safety:

1. Treatment complication in control and intervention groups (SAE-management)
2. A rating committee will provide consistency of the procedure and the assessment of data (e.g. by intraoperative photos, surgery reports, x-rays) to minimize bias

ELIGIBILITY:
Key inclusion criteria:

1. Male or female >30 years of age
2. Lumbar spine pathology with indication for monosegmental PLIF
3. Radiological signs of a degeneration of the adjacent segment without instability

Key exclusion criteria:

1. Radiological signs of existing instability of the adjacent segment 2. Normal endplates and no disc desiccation in MRI in the adjacent seg-ment 3. Previous surgery of the lumbar spine

-

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2011-01; Primary Completion 2012-07 (Estimated); Study Completion 2012-10 (Estimated)

PRIMARY OUTCOMES:
SF36 | 6 Month
  Primary efficacy endpoint:
  The baseline and follow-up values after 6 weeks after the operation as well as 6 and 12 months after baseline of the SF-36 (Short-Form-36)-Measured Outcome regarding the Physical Component Summary (PCS).

SECONDARY OUTCOMES:
1.Mental Component Summary (MCS) and individual dimensions and subscales of the Mental Component Summary (MCS) and individual dimensions and subscales of SF-36 | 6 weeks
  1. Mental Component Summary (MCS) and individual dimensions and subscales of the SF-36 follow-up values after 6 weeks after the operation as well as 6 and 12 months after baseline
Safety | all time
  Assessment of safety:
  1. Treatment complication in control and intervention groups (SAE-management)
  2. A rating committee will provide consistency of the procedure and the assessment of data (e.g. by intraoperative photos, surgery reports, x-rays) to minimize bias
Individual dimensions of the Oswestry Disability Index (ODI) | 6weeks
  Individual dimensions of the Oswestry Disability Index (ODI) follow-up values after 6 weeks after the operation as well as 6 and 12 months after baseline
Time until radiological adjacent instability and comparison to the clinical outcome | 6 weeks
  Time until radiological adjacent instability and comparison to the clinical outcome follow-up values after 6 weeks after the operation as well as 6 and 12 months after baseline
Capacity of work at the time of surgery and after surgery, time until return to work | 6 weeks
  Capacity of work at the time of surgery and after surgery, time until return to work follow-up values after 6 weeks after the operation as well as 6 and 12 months after baseline

CONTACTS AND LOCATIONS:
Overall Officials: Jan Siewe, Dr., Principal Investigator — University of Cologne
Locations (1):
- University of Cologne, Department of Orthopedics& traumasurgery, Cologne, Germany

REFERENCES:
- [Derived] Siewe J, Otto C, Knoell P, Koriller M, Stein G, Kaulhausen T, Eysel P, Zarghooni K, Franklin J, Sobottke R. Comparison of standard fusion with a "topping off" system in lumbar spine surgery: a protocol for a randomized controlled trial. BMC Musculoskelet Disord. 2011 Oct 18;12:239. doi: 10.1186/1471-2474-12-239. PMID 22008088
- See also: Related Info — http://orthopaedie.uk-koeln.de/forschung